CLINICAL TRIAL: NCT01392183
Title: A Randomized Phase 2 Trial of Pazopanib Versus Temsirolimus in Poor-Risk Clear-Cell Renal Cell Carcinoma
Brief Title: Pazopanib Versus Temsirolimus in Poor-Risk Clear-Cell Renal Cell Carcinoma (RCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0358; NCI-2011-01277 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-07-08; First posted 2011-07-12 (Estimated); Results first posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-08

CONDITIONS: Kidney Cancer
Keywords: Kidney cancer; Renal Cell Carcinoma; Poor-Risk Clear-Cell Renal Cell Carcinoma; RCC; Metastatic; Locally advanced; Complete response; CR; Partial Response; PR; Overall survival; OS; Time to progression; TTP; Pazopanib; GW786034; Temsirolimus; CCI-779; Torisel; Benadryl; Diphenhydramine; TemPa
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell; Neoplasm Metastasis; Pathologic Complete Response | interventions — pazopanib; temsirolimus; Surveys and Questionnaires; Diphenhydramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pazopanib (Experimental): Pazopanib 800 mg by mouth daily. Quality of Life Assessment - Completion of full assessment battery at baseline, prior to treatment then every 8 weeks at clinical evaluation.
  Interventions: Drug: Pazopanib; Behavioral: Quality of Life Assessment
- Temsirolimus (Experimental): Temsirolimus 25 mg by vein infused over 30-60 minutes weekly. Benadryl 25 to 50 mg by vein approximately 30 minutes before the start of each dose of temsirolimus. Quality of Life Assessment - Completion of full assessment battery at baseline, prior to treatment then every 8 weeks at clinical evaluation.
  Interventions: Drug: Temsirolimus; Behavioral: Quality of Life Assessment; Drug: Benadryl

INTERVENTIONS:
Drug: Pazopanib — 800 mg by mouth daily in 4 week study cycle.
  Other Names: GW786034
  Arms: Pazopanib
Drug: Temsirolimus — 25 mg by vein infused over 30-60 minutes every week in 4 week study cycle.
  Other Names: CCI-779; Torisel
  Arms: Temsirolimus
Behavioral: Quality of Life Assessment — Completion of full assessment battery at baseline, prior to treatment then every 8 weeks at clinical evaluation.
  Other Names: Questionnaires; Surveys
Drug: Benadryl — 25 to 50 mg by vein approximately 30 minutes before the start of each dose of temsirolimus.
  Other Names: Diphenhydramine
  Arms: Temsirolimus

SUMMARY:
The goal of this clinical research study is to compare pazopanib to temsirolimus in the treatment of advanced clear-cell renal cell carcinoma. The safety of each drug will also be studied.

Pazopanib is designed to block the growth of blood vessels that supply nutrients needed for tumor growth. This may prevent or slow the growth of cancer cells.

Temsirolimus is designed to block the growth of cancer cells, which may cause cancer cells to die.

This is an investigational study. Pazopanib and temsirolimus are both FDA approved and commercially available for the treatment of kidney cancer. It is investigational to compare the 2 drugs.

Up to 90 patients will be enrolled in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
Study Groups and Study Drug Administration:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups. You will have an equal chance of being assigned to either group.

* If you are assigned to Group 1, you will take pazopanib by mouth 1 time every day at about the same time each day on an empty stomach (at least 1 hour before or 2 hours after a meal).
* If you are assigned to Group 2, you will receive temsirolimus by vein 1 time every week over 30-60 minutes. About 30 minutes before you receive each dose of temsirolimus, you will receive Benadryl (diphenhydramine) by vein over 1-2 minutes to help lower the risk of side effects.

If you are assigned to Group 1, do not crush tablets and do not repeat missed doses if it is less than 12 hours until your next scheduled dose. You will be given a pill diary to record when you take each dose. You will return the diary to the study doctor at each study visit.

If you have any side effects, you should tell the study doctor right away. If the study doctor thinks it is in your best interest, your dose may be lowered.

If the disease gets worse while you are on study, you will have the option to change to the study group you were not originally assigned to and take the other study drug. The study drug dosing and study visit schedule will be the same, and the study doctor will discuss any important details with you at the time you change study groups.

Study Visits:

Every 4 weeks on this study is called a study cycle.

Every week during Cycle 1 (Group 1 only), your blood pressure will be checked (either at home, at the clinic, or by your local doctor). If you are checking your own blood pressure at home, you will need to write down your blood pressure in a blood pressure diary each time you check it and bring the diary with you to each clinic visit.

Every 2 weeks for the first 2 cycles (Group 1 only) , blood (about 3 tablespoons) will be drawn for routine tests.

Every week (Group 2 only), blood (about 1 tablespoon) will be drawn for routine tests.

Every cycle (Group 2 only) OR Every other cycle (Group 1 only):

* You will have a physical exam, including measurement of your weight and vital signs.
* You will be asked about any drugs or treatments you may be receiving.
* You will be asked about any side effects you may have had.
* Blood (about 3 tablespoons) will be collected for routine tests.

On Day 1 of Cycle 2, Day 1 of Cycle 4, and every 4 cycles after that (Group 1 only), you will have an ECG to check your heart function.

If you are in Group 2 only, on Day 1 of Cycles 2, 3, and every other cycle after that (Cycles 5, 7, 9, and so on), blood (about 3 tablespoons) will be drawn for routine tests. You will be asked to fast (eat nothing and drink only water) for at least 8 hours before those blood draws.

Every 2 cycles:

* You will have the same imaging scans that you had at screening. After 1 year on treatment, these imaging scans may only be done every 3 cycles (Cycles 5, 8, 11, and so on).
* You will fill out the quality-of-life questionnaires.
* Blood (about 2 teaspoons) will be drawn for tests to check your thyroid function (Group 1 only).
* Urine will be collected for routine tests.

Every 4 cycles, you will have an ECG (Group 2 only).

Every 6 cycles, you will have an ECHO or MUGA scan to check your heart function.

Length of Study:

You may continue taking the study drug for as long as the doctor thinks it is in your best interest. You will no longer be able to take a study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

End-of-Treatment Follow- up:

About 30 days after you stop treatment, during a clinic visit or by phone, you will be asked about any drugs or treatments you may be receiving and any side effects you may have had.

Long-Term Follow-up:

After you stop taking the study drug, the study staff will check up on you to ask how you are doing about every 3 months from then on. The study staff will collect the information they need either from your medical records or by calling you. If you are contacted by phone, the call should only last about 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologic confirmation of metastatic or locally advanced RCC with a major clear cell component.
2. Measurable disease by RECIST criteria.
3. Age >/= 18 years
4. ECOG performance status 0-2 or Karnofsky Performance Status >/= 60%
5. Meets criteria for poor-risk defined as 3 or more of the following: ECOG performance status 2, anemia (hemoglobin lower than reference range), elevated serum LDH > 1.5x upper limit of normal (ULN), hypercalcemia (corrected serum calcium level > upper limit of normal), time from initial RCC diagnosis to registration on this trial < 1 year, and > 1 metastatic organ sites.
6. Adequate organ and marrow function within 14 days of registration as defined below: a) Absolute neutrophil count >/=1,500/µL b) Platelets >/=100,000/µL c) Hgb >/= 9.0 g/dL (transfusion allowed) d) Renal: serum creatinine </= 1.5 x ULN or calculated CrCl >/= 40 cc/min and random urine protein:creatinine ratio (UPC) < 1 or 24-hr urine protein < 1g e) Liver: total bilirubin </= 1.5 mg/dl; AST (SGOT) and ALT (SGPT) </= 2.5 x ULN for subjects without evidence of liver metastases, </= 5 x ULN for subjects with documented liver metastases f) INR </= 1.2 x ULN; PTT </= 1.5 x ULN. Therapeutic anticoagulation with warfarin is allowed if target INR </= 3 on a stable dose of warfarin or on a stable dose of LMW heparin for > 2 weeks (14 days) at time of randomization.
7. Female patients of childbearing potential (not postmenopausal for at least 12 months and not surgically sterile) must have a negative serum or urine pregnancy test within 14 days of study registration. Pregnancy test must be repeated if performed > 14 days before starting study drug.

Exclusion Criteria:

1. Prior malignancy, except for non-melanoma skin cancer, in situ carcinoma of any site, or other cancers for which the patient has been adequately treated and disease free for 2 years
2. Prior targeted therapy (anti-VEGF agents or mTOR inhibitors) including adjuvant therapy, and prior chemotherapy for mRCC. However, prior immunotherapy (cytokines or vaccines) is allowed.
3. Any experimental drug while on this study; however, concomitant bone targeted therapy (bisphosphonates or the anti-RANK ligand denosumab) is allowed.
4. Uncontrolled brain metastases and infections. Patients with brain metastases treated with Gamma Knife (GK) or whole brain radiation within 24 hours of registration.
5. History of stroke within 6 months of registration
6. Clinically significant cardiovascular disease, defined as myocardial infarction (or unstable angina) within 6 months of registration, New York Heart Association (NYHA) Grade II or greater congestive heart failure, serious cardiac dysrhythmia refractory to medical management. However, treated and controlled or stable/not clinically significant cardiovascular disease is allowed per evaluation by cardiologist.
7. Uncontrolled hypertension (home blood pressure readings are permitted) or prior history of hypertensive crisis or hypertensive encephalopathy; however, treatment of hypertension with medications is permitted.
8. History of uncontrolled hemoptysis (>/= 1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1
9. Significant vascular disease including aortic aneurysm, aortic dissection.
10. Symptomatic peripheral vascular disease
11. Pregnancy
12. HIV-positive patients receiving combination anti-retroviral therapy
13. Coagulopathy or bleeding diathesis
14. Concomitant treatment with rifampin, St. John's wort, or the cytochrome p450 enzyme-inducing antiepileptic drugs (phenytoin, carbamazepine or Phenobarbital)
15. Major surgery within 28 days prior to registration
16. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device within 7 days prior to starting drug
17. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study registration
18. Serious non-healing wound
19. Baseline QTcB >/= 470 msec.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2012-10-24 (Actual); Primary Completion 2019-09-08 (Actual); Study Completion 2019-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amado Zurita, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: October 2012 to September 2017
Groups:
- Temsirolimus (Control Group): Temsirolimus 25 mg intravenously weekly. Upon progression patient crosses over over to pazopanib 800 mg orally daily. Treatments stop for progression, toxicity, withdrawal, or death.
- Pazopanib (Treatment Group): Pazopanib 800 mg orally daily. Upon progression patient crosses over to temsirolimus 25 mg intravenously weekly. Treatments stop for progression, toxicity, withdrawal, or death.
Period: First Drug Administration
Arm/Group | Temsirolimus (Control Group) | Pazopanib (Treatment Group)
Started | 35 | 34
Eligible to Cross Over to 2nd Drug (29 participants were eligible to cross over, 8 out of those 29 eligible participants withdrew consent.) | 29 | 31
Completed | 21 | 15
Not Completed | 14 | 19
Not completed — Adverse Event | 3 | 2
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 10 | 17
Period: Second Drug Administration
Arm/Group | Temsirolimus (Control Group) | Pazopanib (Treatment Group)
Started | 21 | 15
Treatment Ended: Progression | 18 | 11
Treatment Ended: Adverse Events | 1 | 2
Treatment Ended: Participant Withdrew | 2 | 1
Treatment Ended: Death | 0 | 1
Completed | 21 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Temsirolimus (Control Group): Temsirolimus 25 mg intravenously weekly. Upon progression patient crosses over to pazopanib 800 mg orally daily. Treatments stop for progression, toxicity, withdrawal, or death.
- Total: Total of all reporting groups
Arm/Group | Temsirolimus (Control Group) | Pazopanib (Treatment Group) | Total
Number analyzed (Participants) | 35 | 34 | 69
Age, Continuous [Median (Full Range); unit: years] | 61 [42 to 80] | 61 [37 to 74] | 61 [37 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 24 | 28 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 11 | 13 | 24
  Unknown or Not Reported | 19 | 18 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 27 | 26 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 35 | 34 | 69
Karnofsky Performance Status (KPS) Score [Count of Participants; unit: Participants] — The KPS score measures the participant's ability to perform ordinary tasks from 100 % - 0%. 100% no signs of disease, 90% minor signs or symptoms of disease, 80% normal activity with effort, 70% cannot do normal daily activities, 60% requires occasional assistance, 50% requires considerable assistance and frequent medical care, 40% disabled requires special care, 30% severely disabled; hospital admission is indicated, 20% very sick; hospital admission needed for active supportive treatment, 10% fatal processes progressing rapidly, and 0% death.
  Participants
    100% | 1 | 1 | 2
    90% | 12 | 10 | 22
    80% | 2 | 2 | 4
    70% | 20 | 21 | 41
Eastern Cooperative Oncology Group (ECOG) Performance Score [Count of Participants; unit: Participants] — ECOG measures how how the disease impacts a participant's daily living abilities such as self-care, daily living activity, and physical ability. The scores ranges from grade 0-5: 0 fully active; 1 restricted in physically strenuous activity but can walk; 2 can walk, capable of all self-care, but cannot do any work activities; 3 capable of only limited self-care and confined to bed or chair more than 50% of waking hours; 4 completely disabled, cannot carry on any self-care, totally confined to bed or chair; and 5 death.
  Participants
    0 | 1 | 1 | 2
    1 | 14 | 12 | 26
    2 | 20 | 21 | 41
Poor -Risk With Disease Eligibility Score. [Count of Participants; unit: Participants] — Participants were considered poor risk with at least 3 factors. The more risk factors the poorer the risk. The factors were any combination of an ECOG grade 2, anemia, high lactate dehydrogenase levels, high calcium levels, less than 1 year from diagnosis to the date of registration on this trial, or more than one organ with metastatic disease.
  Participants
    3 Factors | 12 | 12 | 24
    4 Factors | 18 | 19 | 37
    5 Factors | 5 | 3 | 8
International Metastatic Renal Cell Carcinoma Database Consortium (IMDC) Risk Score [Count of Participants; unit: Participants] — The IMDC score determines the overall survival in participants treated with cancer medications. The score is based on the 6 following factors: less than 1 year from time of diagnosis to trial registration, KPS score of 80% or less, anemia, high levels of calcium, high levels of neutrophils (a type of white blood cell), and a high level of platelets. The scores ranges from 0 - 6. A favorable risk score is 0. An intermediate risk score is 1 - 2. A poor risk score is 3 - 6.
  Participants
    Favorable risk | 0 | 0 | 0
    Intermediate risk | 11 | 8 | 19
    Poor Risk | 24 | 26 | 50

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is measured from the initiation of treatment to the time of first disease progression or death due to any reason during the first drug administration in each arm. Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0), as a 20% or more increase in the sum of the longest diameters of target lesions, or a measurable increase in a non-target lesion or the appearance of new lesions. The PFS median of first drug pazopanib (treatment group) was compared to the PFS median of first drug temsirolimus (control group) in an adjusted Hazard ratio. The hazard ratio compares events from a treatment group to a control group. If the hazard ratio is greater than 1the treatment group performed better. If the hazard ratio is less than 1 the control group performed better. If the hazard ratio is equal to 1, then the groups performed equally.
Time Frame: Measured form start of treatment up to 3 years
Population: The ratio is comparing both arms to each other, therefore the data would be identical.
Measure: Median (Full Range); unit: months
Arm/Group | Temsirolimus (Control Group) | Pazopanib (Treatment Group)
Number analyzed (Participants) | 35 | 34
months | 2.7 [1.2 to 24.6] | 5.2 [0.4 to 34.5]
Statistical Analysis 1: Comparison: Temsirolimus (Control Group) vs Pazopanib (Treatment Group); Test type: Superiority; Hazard Ratio (HR) = 1.36, 95% CI 2-sided [0.84 to 2.22] — Adjusted Hazard Ratio comparing Median PFS of pazopanib (treatment group) to Temsirolimus (control group) as first line of treatment. HR >1 treatment group performed better, < 1 the control group performed better =1 groups performed equally

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is calculated from day of therapy initiation of the first administrated drug to the date of death. Kaplan-Meier estimator used to estimate the OS for each group of participants. The Overall Survival median of first drug pazopanib (treatment group) was compared to the Overall Survival median of first drug temsirolimus (control group) in an adjusted Hazard ratio. The hazard ratio compares events from a treatment group to a control group. If the hazard ratio is greater than 1the treatment group performed better. If the hazard ratio is less than 1 the control group performed better. If the hazard ratio is equal to 1, then the groups performed equally.
Time Frame: From the start of treatment up to 6 years or death, whichever came first
Population: The ratio is comparing both arms to each other, therefore the data would be identical.
Measure: Median (Full Range); unit: months
Groups:
- Pazopanib (Treatment Group): Pazopanib 800 mg orally daily. Pazopanib 800 mg orally daily. Upon progression patient crosses over to temsirolimus 25 mg intravenously weekly. Treatments stop for progression, toxicity, withdrawal, or death
Arm/Group | Temsirolimus (Control Group) | Pazopanib (Treatment Group)
Number analyzed (Participants) | 35 | 34
months | 7.1 [2.4 to 68.8] | 11.9 [1.3 to 63.4]
Statistical Analysis 1: Comparison: Temsirolimus (Control Group) vs Pazopanib (Treatment Group); Test type: Superiority; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.7 to 1.93] — Adjusted HR comparing Median OS of pazopanib (treatment group) to Temsirolimus (control group) as first line of treatment. HR >1 treatment group performed better, < 1 the control group performed better =1 groups performed equally

ADVERSE EVENTS:
Time Frame: Baseline to study completion or date of death from any cause, whichever came first, assessed up to 5 years.
Description: The total at Risk are participants who received the intervention as their first drug or second drug. All participants did not received both drugs.
Arm/Group | Temsirolimus (Control Group) | Pazopanib (Treatment Group)
All-Cause Mortality (participants affected / at risk) | 32/50 | 31/55
Serious Adverse Events (participants affected / at risk) | 15/50 | 10/55
Other Adverse Events (participants affected / at risk) | 35/50 | 33/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temsirolimus (Control Group) (N=50) | Pazopanib (Treatment Group) (N=55)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 2 (2)
Non-cardiac chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chest pain-cardic (Cardiac disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Back Pain (Nervous system disorders) | 0 (0) | 1 (1)
Pain (Nervous system disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Infusion Related Reaction (Immune system disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Platelet Count Decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Creatinine Increased (Renal and urinary disorders) | 1 (1) | 1 (1)
Hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0)
Edema (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Skin breakdown (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temsirolimus (Control Group) (N=50) | Pazopanib (Treatment Group) (N=55)
Abdominal Pain (Gastrointestinal disorders) | 4 (5) | 8 (12)
ALT Increased (Hepatobiliary disorders) | 3 | 19 (47)
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 (10) | 9 (17)
Alk Phos Increased (Hepatobiliary disorders) | 15 (27) | 17 (35)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (8)
Anemia (Blood and lymphatic system disorders) | 31 (112) | 8 (18)
Anorexia (Gastrointestinal disorders) | 9 (15) | 18 (25)
AST increased (Hepatobiliary disorders) | 9 (12) | 19 (53)
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 4 (6)
Chholesterol high (Metabolism and nutrition disorders) | 4 (31) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (8) | 14 (22)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (1)
Creatinine Increased (Renal and urinary disorders) | 20 (34) | 15 (26)
Diarrhea (Gastrointestinal disorders) | 7 (7) | 33 (85)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 3 (3)
Dry Skin (Skin and subcutaneous tissue disorders) | 5 (6) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (13) | 8 (11)
Edema (General disorders) | 18 (45) | 6 (12)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
Fatigue (General disorders) | 5 (9) | 25 (65)
Pain (General disorders) | 4 (6) | 14 (21)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5)
GGT increased (Hepatobiliary disorders) | 0 (0) | 5 (14)
Headache (Nervous system disorders) | 3 (4) | 3 (5)
Hemoglobinuria (Renal and urinary disorders) | 3 (3) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 35 (127) | 22 (38)
Hypernatremia (Metabolism and nutrition disorders) | 2 (5) | 11 (12)
Hypertension (Vascular disorders) | 5 (13) | 26 (53)
Hypertriglyeridemia (Metabolism and nutrition disorders) | 32 (49) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 8 (12) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (5) | 6 (10)
Hyponatremia (Metabolism and nutrition disorders) | 4 (8) | 9 (9)
Hypophosphatemia (Metabolism and nutrition disorders) | 7 (12) | 3 (4)
Hypothyroidism (Endocrine disorders) | 0 (0) | 26 (29)
lymphocyte Count Decreased (Blood and lymphatic system disorders) | 8 (21) | 8 (20)
Mucositis oral (Gastrointestinal disorders) | 27 (48) | 12 (29)
Nausea (Gastrointestinal disorders) | 13 (15) | 32 (79)
Neuropahty (Nervous system disorders) | 1 (1) | 3 (3)
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 (3) | 3 (4)
Palmar-plantar erythrodeysesthesia (Skin and subcutaneous tissue disorders) | 1 (2) | 6 (10)
Parasthesia (Nervous system disorders) | 4 (5) | 5 (9)
Platelet count decreased (Blood and lymphatic system disorders) | 9 (10) | 16 (37)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Proteinuria (Renal and urinary disorders) | 11 (14) | 19 (36)
Rash (Skin and subcutaneous tissue disorders) | 17 (49) | 22 (65)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 20 (38)
Vomiting (Gastrointestinal disorders) | 5 (7) | 23 (44)
Watering eyes (Eye disorders) | 2 (2) | 3 (5)
Weight loss (General disorders) | 4 (4) | 16 (21)
White blood cell decreased (Blood and lymphatic system disorders) | 7 (12) | 10 (24)
Bilirubin increased (Hepatobiliary disorders) | 0 (0) | 6 (11)
Hoarse (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (10)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 9 (12)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 3 (8)
Dysgeusia (Gastrointestinal disorders) | 10 (10) | 19 (26)
Hypoalbuminemia (Investigations) | 4 (5) | 11 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-23): https://cdn.clinicaltrials.gov/large-docs/83/NCT01392183/Prot_SAP_000.pdf